CLINICAL TRIAL: NCT00371943
Title: A Controlled Trial of Ligation Plus Drug Vs. Drug Alone in the Prevention of Variceal Rebleeding
Brief Title: EVL Plus Drug to Prevent Variceal Rebleeding
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: National Science and Technology Council, Taiwan (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EVL
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2006-09-15 (Estimated); Status verified 2006-09

CONDITIONS: Bleeding
Keywords: variceal bleeding,band ligation, beta-blocker; had history of esophageal variceal bleeding
MeSH Terms: conditions — Hemorrhage

INTERVENTIONS:
Procedure: band ligation

SUMMARY:
Both medications with beta-blockers and isosorbide-5-mononitrate and endoscopic variceal ligation have been proven plausible in the prevention of variceal rebleeding. However, the relative efficacy and safety of the combined treatment for preventing rebleeding remains unresolved.

DETAILED DESCRIPTION:
Bleeding from esophageal varices is a severe complication of portal hypertension. After initial control of acute variceal bleeding, patients still carry a high risk of rebleeding. Of those do rebleed, there is a 20%-35% mortality (1). Therefore, preventive procedures are required in patients surviving an episode of acute variceal bleeding. In recent years, endoscopic variceal ligation (EVL) has replaced endoscopic injection sclerotherapy (EIS) as the endoscopic treatment of choice in the management of bleeding esophageal varices (2-3). On the other hand, nonselective beta blockers have been well documented to be effective in reducing variceal rebleeding (4-5). The addition of isosorbide-5-mononitrate (ISMN) has been shown to be even more effective than propranolol alone in the reduction of portal pressure and in the prevention of variceal rebleeding (6). Some studies showed that the combination of nadolol and ISMN is more effective than EIS or EVL in the reduction of variceal rebleeding (7-8). It is still unknown whether EVL combined with nadolol and ISMN is superior to nadolol and ISMN in the prevention of variceal rebleeding. This study was undertaken to compare the effectiveness and complications of ligation plus nadolol and isosorbide mononitrate vs. nadolol plus isosorbide mononitrate for the prevention of variceal rebleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Acute bleeding from esophageal varices (defined below);
2. the etiology of portal hypertension was cirrhosis; and
3. age was between 20 and 75 years old. The diagnosis of cirrhosis was based on pathology, clinical, biochemical, and sonographic or computed tomographic findings. Acute esophageal variceal bleeding was defined as when blood was directly seen by endoscopy to issue from an esophageal varix, or when patients presented with red color signs on their esophageal varices with blood in esophagus or stomach and no other potential site of bleeding identified.

Exclusion Criteria:

1. association with hepatocellular carcinoma or other malignancy,
2. association with cerebral vascular accident, uremia, sepsis or other debilitating disease,
3. had history of gastric variceal bleeding,
4. received beta blocker within one month prior to entry,
5. had history of contraindication to the use of beta blockers, such as asthma, heart failure, atrioventricular block, bradycardia (pulse rate <55/min) or arterial hypotension (systolic blood pressure<90 mmHg).
6. had history of prior shunt operation, TIPS (transjugular intrahepatic portosystemic stent shunt), EIS or EVL,
7. deep jaundice (serum bilirubin >10mg/dl),
8. encephalopathy greater than stage II,
9. failure in control of index variceal bleeding,
10. death within 24 hours of admission, or
11. refused to participate in the trial.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2001-07; Study Completion 2005-03

PRIMARY OUTCOMES:
rebleeding rate

SECONDARY OUTCOMES:
complications

CONTACTS AND LOCATIONS:
Overall Officials: Gin Ho Lo, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Gin-Ho Lo, Kaohsiung City, Taiwan